CLINICAL TRIAL: NCT05948930
Title: Adaptive Working Memory and Physical Exercise Training to Improve Brain and Mitochondrial Function in MCI
Brief Title: Working Memory and Physical Exercise Training in Patients With Mild Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Linda Chang, Principal Investigator, University of Maryland, Baltimore
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HP-00105789
Record Dates: First submitted 2023-07-03; First posted 2023-07-17 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Aerobic Exercise (Experimental): Progressive aerobic exercise 3x/week for 12 weeks.
  Interventions: Behavioral: Progressive aerobic exercise
- Cognitive Training (Experimental): Adaptive cognitive training on Cogmed 5x/week for a total of 25 sessions in 5-8 weeks.
  Interventions: Behavioral: Adaptive cognitive training
- Combined Cognitive and Aerobic Exercise (Experimental): Combined progressive aerobic exercise 3x/week for 12 weeks and adaptive cognitive training on Cogmed 5x/week for a total of 25 sessions in 5-8 weeks simultaneously.
  Interventions: Behavioral: Combined

INTERVENTIONS:
Behavioral: Progressive aerobic exercise — Progressive aerobic exercise
  Arms: Aerobic Exercise
Behavioral: Adaptive cognitive training — Adaptive cognitive training
  Arms: Cognitive Training
Behavioral: Combined — Combine adaptive cognitive and progressive aerobic exercise training
  Arms: Combined Cognitive and Aerobic Exercise

SUMMARY:
The prevalence of dementia will double in the next three decades in the U.S.; effective treatment or prevention for dementia is urgently needed. The current exploratory project aims to evaluate and understand how the brain and cognition may improve after a 12-week intervention that combines brain training and aerobic exercise training to improve brain function, both in those with mild cognitive impairment (some with possible prodromal Alzheimer's disease) and with healthy aging. Findings from this pilot project will guide and refine the development of a future larger clinical trial that aligns with the goals of the National Alzheimer's Plan of Action (NAPA), especially regarding "Prevent and Effectively Treat Alzheimer's Disease (AD) by 2025.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women of all races and ethnicities who are 50-80 years of age will be eligible.
* Only sedentary adults will be eligible (engaging in structured activity for exercise <3x/week) for Progressive aerobic exercise or Combined training
* Ability to use, and accessibility to, an iPad or computer is required for the Adaptive cognitive training and Combined training.
* Fluent in English.
* The diagnosis of MCI will first be confirmed at the screening evaluation using the clinical dementia rating (CDR) scale and the Montreal Cognitive Assessment (MoCA). We will also evaluate their ADL using instrumental activities of daily living (IADL) to ensure they have preserved independence in functional abilities despite the cognitive deficits. The primary caregivers will be interviewed (either in person or by phone) for the participants' IADL to corroborate the independent functional status.

Exclusion Criteria:

* Does not have access to a computer or internet to perform the Cogmed® training AND is unwilling to come to the lab for the training.
* Unable to undergo an MRI investigation based on claustrophobia or metal foreign bodies.
* Symptomatic heart disease, Coronary artery disease, congestive heart failure, uncontrolled hypertension, uncontrolled diabetes (HbA1c>10%), significant cardiovascular disorders (on EKG and graded exercise test) that would prevent the participant from the exercise training; neurologic, musculoskeletal, or other condition that limits the subject's ability to complete study physical assessments.
* Estimated verbal Intelligence Quotient (IQ) below 70 (based on the Wechsler Test of Adult Reading) which would invalidate the informed consent process for the study.
* Self-reported moderate to severe substance use disorder(s) (e.g., self-reported intake >3 oz liquor, or three 4 oz glasses of wine, or three 12 oz cans of beer per day or illicit drug use).
* Severe chronic or acute medical or other (non-MCI) neuropsychiatric conditions that might confound the cognitive or brain imaging measures (e.g., liver function tests >2.5 normal range or evidence for renal failure).
* Body mass index >40 kg/m2.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-01-08 (Actual); Primary Completion 2026-02-07 (Estimated); Study Completion 2026-08-07 (Estimated)

PRIMARY OUTCOMES:
Changes in Brain structure measures | At baseline and at 4 weeks after the corresponding training program.
  Changes in brain volume measures from T1-weighted images (volumes in mm3)
Changes in brain cortical thickness measures | At baseline and at 4 weeks after the corresponding training program.
  Changes in brain cortical thickness measures from T1-weighted images (thickness measures in mm)
Changes in Brain microstructure measures | At baseline and at 4 weeks after the corresponding training program.
  Changes in brain measures of diffused tensor imaging (diffusion coefficient in mm²/s)
Changes in Brain blood flow from Arterial spin labeling magnetic resonance imaging (ASL-MRI) in milliliters/100 g/minutes | At baseline and at 4 weeks after the corresponding training program.
  Changes in Brain blood flow from Arterial spin labeling magnetic resonance imaging (ASL-MRI) in milliliters/ 100 g/ minutes
Changes in Brain Activation on functional MRI | At baseline and at 4 weeks after the corresponding training program.
  Changes in functional MRI from blood oxygen level dependence (BOLD) contrast on fMRI (in percentage change)
Changes in cognitive performance, emotions, and motor function based on NIH toolbox | At baseline and at 4 weeks after the corresponding training program.
  Changes in cognitive performance, emotions, and motor function in raw scores measured by the NIH Toolbox® (reports will be generated as T scores, with higher T scores indicating better outcomes)
Changes in executive function using the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) | At baseline and at 4 weeks after the corresponding training program.
  Changes in executive function using the Behavior Rating Inventory of Executive Function-Adult Version (BRIEF-A) (reports will be generated as T scores, with lower T scores indicating better outcomes and T scores higher than 65 indicating significant impairments in the executive function)
Changes in Blood Bioenergetic Markers | At baseline and at 4 weeks after the corresponding training program.
  Platelet mitochondrial respiration (OCR) and extracellular acidification rates (ECAR) will be evaluated to assess bioenergetic profiles in platelets isolated from whole blood of fasted participants. OCR will be measured using a Seahorse model XFe96 machine as the high throughput platform. Measurements of OCR/ECAR will be performed with the following modifications. Platelets will be isolated from whole blood with a Beckman Allegra model X-30R centrifuge.
  Platelets will be counted using a Nexcelom Bioscience Cellometer (Lawrence, MA) using Calcein acetoxymethyl (AM) ester dye to enable the seeding of 10,000,000 platelets per well.

SECONDARY OUTCOMES:
VO2peak | At baseline and within one week after the corresponding training program.
  VO2peak will be used as the primary measure of aerobic capacity. Subjects will be asked to exercise to voluntary exhaustion during a treadmill test using a modified Bruce protocol. Oxygen (O2) consumption, carbon dioxide (CO2) production, and minute ventilation will be measured breath-by-breath using a metabolic cart and the average of the final two 20 second values of O2 consumption are VO2peak.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Baltimore, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chacko BK, Kramer PA, Ravi S, Benavides GA, Mitchell T, Dranka BP, Ferrick D, Singal AK, Ballinger SW, Bailey SM, Hardy RW, Zhang J, Zhi D, Darley-Usmar VM. The Bioenergetic Health Index: a new concept in mitochondrial translational research. Clin Sci (Lond). 2014 Sep;127(6):367-73. doi: 10.1042/CS20140101. PMID 24895057
- [Background] Vidorreta M, Wang Z, Chang YV, Wolk DA, Fernandez-Seara MA, Detre JA. Whole-brain background-suppressed pCASL MRI with 1D-accelerated 3D RARE Stack-Of-Spirals readout. PLoS One. 2017 Aug 24;12(8):e0183762. doi: 10.1371/journal.pone.0183762. eCollection 2017. PMID 28837640
- [Background] Dolui S, Vidorreta M, Wang Z, Nasrallah IM, Alavi A, Wolk DA, Detre JA. Comparison of PASL, PCASL, and background-suppressed 3D PCASL in mild cognitive impairment. Hum Brain Mapp. 2017 Oct;38(10):5260-5273. doi: 10.1002/hbm.23732. Epub 2017 Jul 24. PMID 28737289
- [Background] Hol HR, Flak MM, Chang L, Lohaugen GCC, Bjuland KJ, Rimol LM, Engvig A, Skranes J, Ernst T, Madsen BO, Hernes SS. Cortical Thickness Changes After Computerized Working Memory Training in Patients With Mild Cognitive Impairment. Front Aging Neurosci. 2022 Apr 4;14:796110. doi: 10.3389/fnagi.2022.796110. eCollection 2022. PMID 35444526
- [Background] Panee J, Gerschenson M, Chang L. Associations Between Microbiota, Mitochondrial Function, and Cognition in Chronic Marijuana Users. J Neuroimmune Pharmacol. 2018 Mar;13(1):113-122. doi: 10.1007/s11481-017-9767-0. Epub 2017 Nov 4. PMID 29101632
- [Background] Tyrrell DJ, Bharadwaj MS, Jorgensen MJ, Register TC, Shively C, Andrews RN, Neth B, Keene CD, Mintz A, Craft S, Molina AJA. Blood-Based Bioenergetic Profiling Reflects Differences in Brain Bioenergetics and Metabolism. Oxid Med Cell Longev. 2017;2017:7317251. doi: 10.1155/2017/7317251. Epub 2017 Oct 2. PMID 29098063
- [Background] Chang L, Holt JL, Yakupov R, Jiang CS, Ernst T. Lower cognitive reserve in the aging human immunodeficiency virus-infected brain. Neurobiol Aging. 2013 Apr;34(4):1240-53. doi: 10.1016/j.neurobiolaging.2012.10.012. Epub 2012 Nov 15. PMID 23158761
- [Background] Chang L, Yakupov R, Cloak C, Ernst T. Marijuana use is associated with a reorganized visual-attention network and cerebellar hypoactivation. Brain. 2006 May;129(Pt 5):1096-112. doi: 10.1093/brain/awl064. Epub 2006 Apr 3. PMID 16585053
- [Background] Tomasi D, Caparelli EC, Chang L, Ernst T. fMRI-acoustic noise alters brain activation during working memory tasks. Neuroimage. 2005 Aug 15;27(2):377-86. doi: 10.1016/j.neuroimage.2005.04.010. PMID 15893942
- [Background] Tomasi D, Ernst T, Caparelli EC, Chang L. Practice-induced changes of brain function during visual attention: a parametric fMRI study at 4 Tesla. Neuroimage. 2004 Dec;23(4):1414-21. doi: 10.1016/j.neuroimage.2004.07.065. PMID 15589105
- [Background] Ernst T, Chang L, Arnold S. Increased glial metabolites predict increased working memory network activation in HIV brain injury. Neuroimage. 2003 Aug;19(4):1686-93. doi: 10.1016/s1053-8119(03)00232-5. PMID 12948723
- [Background] Ernst T, Chang L, Jovicich J, Ames N, Arnold S. Abnormal brain activation on functional MRI in cognitively asymptomatic HIV patients. Neurology. 2002 Nov 12;59(9):1343-9. doi: 10.1212/01.wnl.0000031811.45569.b0. PMID 12427881
- [Background] Chang L, Lohaugen GC, Douet V, Miller EN, Skranes J, Ernst T. Neural correlates of working memory training in HIV patients: study protocol for a randomized controlled trial. Trials. 2016 Feb 2;17:62. doi: 10.1186/s13063-016-1160-4. PMID 26833223
- [Background] Flak MM, Hernes SS, Chang L, Ernst T, Douet V, Skranes J, Lohaugen GC. The Memory Aid study: protocol for a randomized controlled clinical trial evaluating the effect of computer-based working memory training in elderly patients with mild cognitive impairment (MCI). Trials. 2014 May 3;15:156. doi: 10.1186/1745-6215-15-156. PMID 24886034
- [Background] Chang L, Lohaugen GC, Andres T, Jiang CS, Douet V, Tanizaki N, Walker C, Castillo D, Lim A, Skranes J, Otoshi C, Miller EN, Ernst TM. Adaptive working memory training improved brain function in human immunodeficiency virus-seropositive patients. Ann Neurol. 2017 Jan;81(1):17-34. doi: 10.1002/ana.24805. Epub 2016 Dec 28. PMID 27761943
- [Background] Brehmer Y, Westerberg H, Backman L. Working-memory training in younger and older adults: training gains, transfer, and maintenance. Front Hum Neurosci. 2012 Mar 27;6:63. doi: 10.3389/fnhum.2012.00063. eCollection 2012. PMID 22470330
- [Background] Kramer AF, Colcombe S. Fitness Effects on the Cognitive Function of Older Adults: A Meta-Analytic Study-Revisited. Perspect Psychol Sci. 2018 Mar;13(2):213-217. doi: 10.1177/1745691617707316. PMID 29592650
- [Background] Kramer AF, Erickson KI. Capitalizing on cortical plasticity: influence of physical activity on cognition and brain function. Trends Cogn Sci. 2007 Aug;11(8):342-8. doi: 10.1016/j.tics.2007.06.009. Epub 2007 Jul 12. PMID 17629545